CLINICAL TRIAL: NCT06037096
Title: Implementation of a Structured Post-pulmonary Embolism Follow-up Model in a Danish Hospital Setting
Brief Title: Implementation of a Structured Post-pulmonary Embolism Follow-up Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Stine Foged Lindegaard, PhD student, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Attend-PE
Record Dates: First submitted 2023-06-20; First posted 2023-09-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism
Keywords: Implementation; Health related quality of life; Intervention; Pulmonary embolism; Health care model
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Attend-PE (Experimental)
  Interventions: Other: Attend-PE model

INTERVENTIONS:
Other: Attend-PE model — A pulmonary embolism follow-up care model consisting of structured elements for follow-up after discharge from hospital.
  Other Names: A structured post-pulmonary embolism follow-up model

SUMMARY:
Venous thromboembolism (VTE), clinically presenting as deep vein thrombosis or pulmonary embolism (PE) is the third most frequent cardiovascular disease and is associated with substantial short- and long-term morbidity and mortality and high costs of care. In addition negative physical and mental complications following VTE are common. However in terms of PE, there are no structured follow-up programs in Denmark and there is considerable variation in practice patterns of post-PE management both within and between countries.

This project aims to develop, test and implement a structured follow-up care model for patients with PE (The Attend-PE model). This project is a pre-post intervention study and will estimate the effectiveness of implementing the structured follow-up care model on a national level.

DETAILED DESCRIPTION:
The pre-post intervention study aims to measure differences in self-reported and clinical outcomes in patients with PE before and after the developed Attend-PE model has been implemented.

For the pre-intervention period, patient-reported questionnaires and registry data will be collected on all persons having received a CT-verified diagnosis of PE in the period March 2022 - May 2023. At 6 and 12 months following the PE event, the patients will receive an online letter with an invitation to complete an online questionnaire. The questionnaire includes validated patient-reported outcome measures and questions about sociodemographic factors. Furthermore, for all patients who have been invited to participate, register data will be retrieved on use of health care services, sick leave, prescription medication, as well as information on hospital of admission. Thus, the last PROM and register data for the 12-month follow-up will be retrieved in May 2024.

From October 2023 - Juni 2024 implementation of the Attend-PE model takes place on a national level, with a project team managing training of personnel and supporting the reorganization of care at the participating hospitals. 16 Danish hospitals have agreed to participate.

Following the implementation of the Attend-PE model, the post-intervention period is initiated. From October 2023 - Juni 2025 a data collection period similar to the pre-intervention period will take place, with patient-reported questionnaires forwarded to patients following a diagnosis of PE at 6 and 12 months, and data from registries being collected in the same time period. Thus, the last 12-month follow-up is expected to be completed in Juni 2026.

Detailed description of Attend-PE model:

* During hospitalization patients are given standardized patient information. This includes a written leaflet, oral information and links for online information (e.g., videos). An assessment of need for cancer screening is made, and in case of symptomatic DVT compressions stockings are provided. Before discharge patients are referred to a VTE clinic.
* Following discharge, patients and their relatives are invited to participate in a 2-hour group-based patient education session, ideally taking place within the first 2 weeks after discharge. This is managed by a nurse, physician and/or allied health professional and includes education about the condition, treatment, symptom management, physical and mental health, importance of physical activity and social support, and an overview of the care pathway. Time is given for questions and discussion with peers.
* Following the patient education, an individual follow-up consultation is offered, depending on an assessment of the individual patients needs. This allows for a recapitulation of the previous information given, and specific questions or worries related to the individual patients situation.
* At three months post-discharge, patients are invited for a consultation with a physician at the VTE clinic. Prior to the consultation, the patient completes an online questionnaire in the waiting room, including validated questionnaires about treatment satisfaction (Anti-Clot Treatment Scale) and physical and mental wellbeing (Pulmonary Embolism Quality of Life with cascading questions about dyspnea (MRC), anxiety (GAD-7) and depression (PHQ-9). The physician uses the patients responses actively during the consultation for discussion of continued treatment and assessment of whether further referral is required, i.e. to physiotherapist for assessment of physical function and rehabilitation needs, or to the GP for assessment of anxiety or depression and potential treatment hereof. If CTEPH is suspected, referral for VQ scan and/or echochardiography is made. Finally, referral for genetic testing may be considered if thrombophilia is suspected. For patients with provoked PE where medical treatment is completed at 3 months, and where none of the above referrals are required, patients are referred to their GP with standardized a discharge summary for the GP, and information material for the patient.
* For patients continuing medical treatment, a new consultation with a nurse is planned at 6 months, depending on the patients needs. Core elements are adjustment of medication and assessment of physical and psychosocial well-being.
* For patients with individual needs due to complex health conditions, frailty, few psychosocial resources or similar, extra consultations may be provided during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years)
* CT-verified diagnosis of PE

Exclusion Criteria:

* patients who are not living in Denmark on the extraction date
* patients with a active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The Pulmonary Embolism Quality of Life (PEmb-QoL) questionnaire | 6 and 12 month follow-up
  42 item covering health-related quality of life after pulmonary embolism. Transformed scale show score from 0-100, where 0 is the worst outcome and 100 is the best outcome.
Adherence to the anticoagulant treatment | within the first 6 and 12 months
  Patients having redeemed ≥80% of the prescribed anticoagulant medication. Using The Danish National Prescription Registry.

SECONDARY OUTCOMES:
EuroQol 5 Dimensions (EQ-5D) | 6 and 12 month follow-up
  Covering general Health in five dimension. The scores fall on a scale of -0.757 (worst health state) to 1.0 (best health state).
Post-VTE Functional Status Scale (PFVS) | 6 and 12 month follow-up
  Covering functional status in 5 categories of functional limitations. In total 5 grades of functional limitations, where 1 is the worst grade and 5 is the best grade.
Anti-Clot Treatment Scale (ACTS) | 6 and 12 month follow-up
  Covering satisfaction with anticoagulant treatment (12-item ACTS Burdens scale and 3-item ACTS Benefits scale). 5-point to 7-point scales, where higher scores indicate higher satisfaction with treatment.
General Anxiety Disorder-7 (GAD7) | 6 and 12 month follow-up
  Covering anxiety. Score from 0-3 and total score range from 0 to 21, where 21 is the worst outcome and 0 is the best outcome.
Patient Health Questionnaire (PHQ-9) | 6 and 12 month follow-up
  Covering depression. Score from 0-3 and total score range from 0 to 27, where 27 is the worst outcome and 0 is the best outcome.
Patient Activation Measure (PAM) | 6 and 12 month follow-up
  Covering individual's knowledge, skills and confidence integral to managing one's own health and healthcare on a 4-point likert scale. Transformed scale show score from 0-100, where 0 is the worst outcome and 100 is the best outcome.
Work Productivity and Activity Impairment questionnaire (WPAI:GH, v2.0.) | 6 and 12 month follow-up
  Covering work productivity and activity impairment (6 questions). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Recurrent VTE | within the first 6 and 12 months
  New hospital admission with a diagnosis of deep vein thrombosis or pulmonary embolism. Using the Danish National Patient registry (DNPR).
Major and clinically relevant nonmajor bleeding | within the first 6 and 12 months
  According to The International Society for Thrombosis and Haemostasis (ISTH) definitions. Using the Danish National Patient registry (DNPR).
VTE-related death | within the first 6 and 12 months
  Death of VTE. Using the Danish Death Register and CPR Registry.

CONTACTS AND LOCATIONS:
Overall Officials: Anette A. Højen, Principal Investigator — Aalborg University Hospital; Nanna Rolving, Principal Investigator — Aarhus University Hospital; Søren P. Johnsen, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindegaard SF, Hojen AA, Rolving N. Electronic adaptation and danish cross-cultural translation of PEmb-QoL and VEINES-QoL/Sym for patients with venous thromboembolism. J Patient Rep Outcomes. 2024 Feb 26;8(1):21. doi: 10.1186/s41687-024-00698-9. PMID 38407682
- [Background] Rolving N, Lindegaard SF, Johnsen SP, Grove EL, Kumler T, Valentin JB, Risor BW, Klok FA, Konstantinides S, Hojen AA. Effectiveness and cost-effectiveness of a structured integrated post-pulmonary embolism follow-up care model (Attend-PE): a rationale and protocol for a multicentre clinical pre-post study. BMJ Open. 2024 Dec 11;14(12):e088533. doi: 10.1136/bmjopen-2024-088533. PMID 39663161
- [Background] Hojen AA, Lindegaard SF, Grove EL, Hansen AL, Larsen TB, Kumler T, Johnsen SP, Rolving N. Development of A structured integrated post-Pulmonary Embolism care model: The Attend-PE model. J Thromb Haemost. 2024 Nov;22(11):3137-3147. doi: 10.1016/j.jtha.2024.06.027. Epub 2024 Aug 8. PMID 39122195
- [Background] Hansen AL, Hojen AA, Lindegaard SF, Grove EL, Jakobsen C, Rolving N. The Attend-PE model: A feasibility study of a structured follow-up care model for patients with pulmonary embolism. Thromb Res. 2024 Oct;242:109133. doi: 10.1016/j.thromres.2024.109133. Epub 2024 Aug 24. PMID 39216272